CLINICAL TRIAL: NCT03137238
Title: Optic Flow and Vestibular Sensory Integration in Self-motion Perception in Parkinson's Disease
Brief Title: Self-motion Perception in Parkinson's Disease
Acronym: SMP_PD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Bar-Ilan University, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: SHEBA-16-3707-SDIK-CTIL
Record Dates: First submitted 2017-04-18; First posted 2017-05-02 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2020-03

CONDITIONS: Parkinson Disease
Keywords: Self-motion perception; Optic flow; Vestibular system; Multisensory integration; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Early_PD: People with Parkinson's disease in the early stages with low doses of antiparkinsonian medication and no motor fluctuations.
  Interventions: Other: Investigation of self-perception in Parkinson's disease
- Advanced_PD: People with advanced Parkinson's disease with motor fluctuations.
  Interventions: Other: Investigation of self-perception in Parkinson's disease
- Early_controls: Healthy participants matched for age and gender to the 'Early_PD' group.
  Interventions: Other: Investigation of self-perception in Parkinson's disease
- Advanced_controls: Healthy participants matched for age and gender to the 'Advanced_PD' group.
  Interventions: Other: Investigation of self-perception in Parkinson's disease

INTERVENTIONS:
Other: Investigation of self-perception in Parkinson's disease — There is no therapeutic intervention.

SUMMARY:
Parkinson's Disease as well as being a disorder of motor function also causes a wide range of non-motor disturbances many of which are involved in the prodromal stage prior to the onset of motor symptoms. Abnormal perception in the visual and in other domains is increasingly being recognized. Control of the movement of our bodies in space involves perception of self-motion which is dependent on the processing and integration of multimodality information from the kinesthetic, proprioceptive, visual (mostly optic flow) and vestibular systems. Dysfunction in this process may contribute to disturbed postural control and thus result in gait abnormalities and falls which are common as Parkinson's disease progresses, is difficult to treat and causes disability and a loss of independence.

The integration of information from different modalities ("multisensory integration") is vital for intact perception of the world. Theoretical studies, based on Bayesian statistics, have provided a framework to study multisensory-integration with predictions for an 'optimal' strategy.

Many human and animal studies have demonstrated near optimal cue-integration. Yet, while multisensory integration is an active topic of research in normal brain function, with well-established tools, it has not been studied in PD. The investigators hypothesize, based on the apparent over-dependence in PD on visual cues that PD patients will demonstrate defective multisensory integration. This can have profound effects on basic motor functions. Furthermore, based on both visual and vestibular abnormalities (described above) the basic (uni-sensory) performance may also be degraded in PD.

In this study the investigators will observe the basic (uni-sensory) and the multisensory integration of visual and vestibular perception of self-motion within the same experiment.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is classically characterized by a decline in motor function, marked by the hallmark symptoms of akinesia, bradykinesia, rigidity and tremor as well as impaired posture and balance. However, non-motor symptoms are also recently becoming recognized as a major part of the disease. Non-motor symptoms may include sleep disorders, mood disturbances, hallucinations, cognitive impairment, and various sensory and perceptual deficits. In contrast to the motor symptoms, non-motor symptoms are less observable by nature, and can therefore go unnoticed if not tested directly.

Already, early studies revealed broad visual dysfunction in PD. This includes delays in visual evoked responses and abnormalities in contrast, spatiotemporal and color sensitivity. PD patients also have altered perception of visual orientation as well as complex visual impairments. Yet, despite their visual deficits, PD patients seem to be functionally more dependent on vision, versus controls. This seems to contradict established principles of optimal sensory integration, according to which, impaired cues should be less relied upon. However, this can only be gauged within a principled framework that measures, quantifies and compares the precision of relevant perceptual cues. Namely, it is the relative reliabilities of sensory cues that should, according to schemes of optimal (Bayesian) integration, set the extent to which the cues are relied upon (related to further below).

Research has demonstrated impairments in sensory systems, other than vision, such as proprioceptive and vestibular function. Interestingly, many sensory deficits in PD may be closely associated with "classic" motor symptoms. For example: : i) dysfunctional vestibular signals may lead to impaired balance control in PD, (ii) proprioceptive deficits impair voluntary and reflexive motor commands, (iii) impairments in spatial perception may contribute to freezing of gait (FOG), and (iv) PD patients overestimate the volume of their own speech, likely reflecting perceptual deficits either by impaired sensorimotor integration or by impaired self-awareness of motor deficits. Also, higher perceptual functions, such as perception of emotion from facial expression, is impaired in parkinsonian patients. Perception of self-motion arises primarily from inertial motion (vestibular) and optic flow (visual) cues. When presented with radial expanding optic flow patterns, PD patients demonstrate altered navigational veering and altered perception of the egocentric midline as well as reduced activation in visual brain areas versus controls. However, thresholds of self-motion perception from optic flow have not yet been investigated, and will thus be measured in this study.

Vestibular abnormalities might also affect perception of self-motion in PD. Recently, Bertolini et al. (2015) found impaired tilt perception in PD, but here too, vestibular thresholds of linear self-motion perception have not been researched directly. Hence, the first aim of this study is to determine the thresholds of unisensory (visual and vestibular) perception of self-motion in PD, using a rigorous and well used paradigm of heading discrimination.

However, in addition to deficits in visual and vestibular perception of self-motion, PD patients may suffer from sub-optimal integration of these cues. Hence, the second major aim is to specifically investigate the integration of visual and vestibular cues for self-motion perception. This will be done in the Bayesian framework of multisensory integration.

The integration of information from different modalities ("multisensory integration") is vital for intact perception of the world. Theoretical studies, based on Bayesian statistics, have provided a framework to study multisensory-integration with predictions for an 'optimal' strategy. Assuming Gaussian distribution and a flat prior, optimal integration of multiple cues reduces to straight forward linear equation, according to which the multisensory percept is a weighted combination of the underlying cues. Many human and animal studies have indeed demonstrated near optimal cue-integration. Yet, while multisensory integration is an active topic of research in normal brain function, with well-established tools, it has not been studied in PD.The investigators hypothesize, based on the apparent over-dependence in PD on visual cues. PD patients might demonstrate non-optimal multisensory integration (namely overweighting of visual cues). This can have profound effects on basic function.

Adding sensory noise to a stimulus reduces its reliability. In the optic flow stimuli of self-motion through a 3D cloud of dots, reliability can be controlled by manipulating the coherence of the moving dots. For 100% coherence (no added noise), all the dots move coherently according to the direction of simulated self-motion. When noise is added, e.g. to 75% coherence, 75% of the dots move coherently according to the direction of self-motion, whereas the remaining 25% move in a random direction As coherence is decreased the visual stimulus reliability reduces. Recently the investigators showed that different clinical groups (e.g. autism) can respond differently to the addition of visual noise. Hence, as part of these experiments, the investigators will also compare visual perception in the absence and presence of added visual noise. The pathophysiology of PD is often understood to reflect increased neuronal noise (e.g. beta oscillations) hence the investigators hypothesize that external sensory noise might have a stronger effect on PD patients vs. controls (perhaps by the stimulus aggravating, rather than reducing, neuronal fluctuations in PD).

Hence, in this study the investigators have 3 main aims: i) to observe the basic (unisensory) visual and vestibular perception of self-motion in PD, ii) to observe the multisensory integration in PD patients, within the framework of Bayesian inference, and iii) to observe the effects of reducing visual reliability (the addition of visual stimulus noise) on performance in PD. All three aims will be addressed with the same experiment. All participants will come for two visits. PD patients will perform the same procedure once "on" medication and once "off" medication (the order of which will be counterbalanced between patients; determined randomly in advance). For the "off" medication condition, patients will stop taking their PD medication 12 hours before the experiments (until after the experiment). The control group will also perform the experiment twice in order to control the possible artifact of learning effects.

ELIGIBILITY:
Inclusion Criteria:

* Both groups will be screened using the Montreal Cognitive Assessment (MoCA) test, and only individuals with normal cognitive function will be included in the study (above 22)

Exclusion Criteria:

* PD patients determined clinically to be at high risk of falling, indicated by scores of 3 or more on items 2.12, 2.13, 3.10, 3.11 and 3.12 of the Movement Disorder Society- Unified Parkinson's Disease Rating Scale (MDS- UPDRS).
* Participants under 18 years old
* Participants with vertigo or other active vestibular disease

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PD patients and healthy subjects.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change in multisensory integration | All participants will come for two visits, each visit will take 1.5 - 2 hours 4 days and two weeks apart. Measurements will be taken in a continuous fashion during these visits only.
  Psychometric plot will be defined as the proportion of rightward choices as a function of heading angle and calculated by fitting the data with a cumulative Gaussian distribution function. Separate psychometric functions will construct for visual, vestibular, and combined cues. The psychophysical threshold and point of subjective equality will be the SD (σ) and mean (μ), respectively, deduced from the fitted distribution function. We will compare the actual weights patients gave to each cue to the predicted one, and thus will be able to study if their integration was optimal, compere to healthy participants. No change is expected to occur for control group. For the PD group, there may be an effect of antiparkinsonian medications, hence PD participants will be tested once after taking the regular antiparkinsonian medications and once after a 12 hour period of not taking any antiparkinsonian medication.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Israeli-Korn, Dr, Principal Investigator — Institute of Movement Disorders, Sheba medical center, Tel-Hashomer; Adam Zaidel, PhD, Principal Investigator — Gonda Multidisciplinary Brain Research Center at Bar-Ilan University, Ramat-Gan
Locations (2):
- Israel (2):
  - Sheba Medical Center, Ramat Gan
  - Bar Ilan University, Ramat Gan

IPD SHARING:
Plan to Share IPD: No
There is currently no plan for sharing IPD

REFERENCES:
- [Background] Almeida QJ, Lebold CA. Freezing of gait in Parkinson's disease: a perceptual cause for a motor impairment? J Neurol Neurosurg Psychiatry. 2010 May;81(5):513-8. doi: 10.1136/jnnp.2008.160580. Epub 2009 Sep 15. PMID 19758982
- [Background] Azulay JP, Mesure S, Amblard B, Pouget J. Increased visual dependence in Parkinson's disease. Percept Mot Skills. 2002 Dec;95(3 Pt 2):1106-14. doi: 10.2466/pms.2002.95.3f.1106. PMID 12578250
- [Background] Ho AK, Bradshaw JL, Iansek T. Volume perception in parkinsonian speech. Mov Disord. 2000 Nov;15(6):1125-31. doi: 10.1002/1531-8257(200011)15:63.0.co;2-r. PMID 11104195
- [Background] Davidsdottir S, Wagenaar R, Young D, Cronin-Golomb A. Impact of optic flow perception and egocentric coordinates on veering in Parkinson's disease. Brain. 2008 Nov;131(Pt 11):2882-93. doi: 10.1093/brain/awn237. Epub 2008 Oct 28. PMID 18957454
- [Background] Fetsch CR, Turner AH, DeAngelis GC, Angelaki DE. Dynamic reweighting of visual and vestibular cues during self-motion perception. J Neurosci. 2009 Dec 9;29(49):15601-12. doi: 10.1523/JNEUROSCI.2574-09.2009. PMID 20007484
- [Background] Gu Y, Angelaki DE, Deangelis GC. Neural correlates of multisensory cue integration in macaque MSTd. Nat Neurosci. 2008 Oct;11(10):1201-10. doi: 10.1038/nn.2191. Epub 2008 Sep 7. PMID 18776893
- [Background] Gullett JM, Price CC, Nguyen P, Okun MS, Bauer RM, Bowers D. Reliability of three Benton Judgment of Line Orientation short forms in idiopathic Parkinson's disease. Clin Neuropsychol. 2013;27(7):1167-78. doi: 10.1080/13854046.2013.827744. Epub 2013 Aug 19. PMID 23957375
- [Background] Zaidel A, Goin-Kochel RP, Angelaki DE. Self-motion perception in autism is compromised by visual noise but integrated optimally across multiple senses. Proc Natl Acad Sci U S A. 2015 May 19;112(20):6461-6. doi: 10.1073/pnas.1506582112. Epub 2015 May 4. PMID 25941373
- [Background] Zaidel A, Spivak A, Grieb B, Bergman H, Israel Z. Subthalamic span of beta oscillations predicts deep brain stimulation efficacy for patients with Parkinson's disease. Brain. 2010 Jul;133(Pt 7):2007-21. doi: 10.1093/brain/awq144. Epub 2010 Jun 9. PMID 20534648
- [Background] Weil RS, Schrag AE, Warren JD, Crutch SJ, Lees AJ, Morris HR. Visual dysfunction in Parkinson's disease. Brain. 2016 Nov 1;139(11):2827-2843. doi: 10.1093/brain/aww175. PMID 27412389
- [Background] Postuma RB, Berg D, Stern M, Poewe W, Olanow CW, Oertel W, Obeso J, Marek K, Litvan I, Lang AE, Halliday G, Goetz CG, Gasser T, Dubois B, Chan P, Bloem BR, Adler CH, Deuschl G. MDS clinical diagnostic criteria for Parkinson's disease. Mov Disord. 2015 Oct;30(12):1591-601. doi: 10.1002/mds.26424. PMID 26474316
- [Background] Montse A, Pere V, Carme J, Francesc V, Eduardo T. Visuospatial deficits in Parkinson's disease assessed by judgment of line orientation test: error analyses and practice effects. J Clin Exp Neuropsychol. 2001 Oct;23(5):592-8. doi: 10.1076/jcen.23.5.592.1248. PMID 11778636
- [Background] Morgan ML, Deangelis GC, Angelaki DE. Multisensory integration in macaque visual cortex depends on cue reliability. Neuron. 2008 Aug 28;59(4):662-73. doi: 10.1016/j.neuron.2008.06.024. PMID 18760701
- [Background] Stein BE, Stanford TR. Multisensory integration: current issues from the perspective of the single neuron. Nat Rev Neurosci. 2008 Apr;9(4):255-66. doi: 10.1038/nrn2331. PMID 18354398
- [Background] Revonsuo A, Portin R, Koivikko L, Rinne JO, Rinne UK. Slowing of information processing in Parkinson's disease. Brain Cogn. 1993 Jan;21(1):87-110. doi: 10.1006/brcg.1993.1007. PMID 8424865
- [Background] Sprengelmeyer R, Young AW, Mahn K, Schroeder U, Woitalla D, Buttner T, Kuhn W, Przuntek H. Facial expression recognition in people with medicated and unmedicated Parkinson's disease. Neuropsychologia. 2003;41(8):1047-57. doi: 10.1016/s0028-3932(02)00295-6. PMID 12667540
- [Background] van der Hoorn A, Renken RJ, Leenders KL, de Jong BM. Parkinson-related changes of activation in visuomotor brain regions during perceived forward self-motion. PLoS One. 2014 Apr 22;9(4):e95861. doi: 10.1371/journal.pone.0095861. eCollection 2014. PMID 24755754
- [Background] Ricciardi L, Visco-Comandini F, Erro R, Morgante F, Bologna M, Fasano A, Ricciardi D, Edwards MJ, Kilner J. Facial Emotion Recognition and Expression in Parkinson's Disease: An Emotional Mirror Mechanism? PLoS One. 2017 Jan 9;12(1):e0169110. doi: 10.1371/journal.pone.0169110. eCollection 2017. PMID 28068393
- [Background] Knill DC, Pouget A. The Bayesian brain: the role of uncertainty in neural coding and computation. Trends Neurosci. 2004 Dec;27(12):712-9. doi: 10.1016/j.tins.2004.10.007. PMID 15541511
- [Background] Konczak J, Corcos DM, Horak F, Poizner H, Shapiro M, Tuite P, Volkmann J, Maschke M. Proprioception and motor control in Parkinson's disease. J Mot Behav. 2009 Nov;41(6):543-52. doi: 10.3200/35-09-002. PMID 19592360
- [Background] Bertolini G, Wicki A, Baumann CR, Straumann D, Palla A. Impaired tilt perception in Parkinson's disease: a central vestibular integration failure. PLoS One. 2015 Apr 15;10(4):e0124253. doi: 10.1371/journal.pone.0124253. eCollection 2015. PMID 25874868
- [Background] Bodis-Wollner I, Yahr MD. Measurements of visual evoked potentials in Parkinson's disease. Brain. 1978 Dec;101(4):661-71. doi: 10.1093/brain/101.4.661. PMID 737524
- [Background] Bodis-Wollner I, Marx MS, Mitra S, Bobak P, Mylin L, Yahr M. Visual dysfunction in Parkinson's disease. Loss in spatiotemporal contrast sensitivity. Brain. 1987 Dec;110 ( Pt 6):1675-98. doi: 10.1093/brain/110.6.1675. PMID 3427405
- [Background] Fushiki H, Kobayashi K, Asai M, Watanabe Y. Influence of visually induced self-motion on postural stability. Acta Otolaryngol. 2005 Jan;125(1):60-4. doi: 10.1080/00016480410015794. PMID 15799576
- [Background] Maier F, Prigatano GP, Kalbe E, Barbe MT, Eggers C, Lewis CJ, Burns RS, Morrone-Strupinsky J, Moguel-Cobos G, Fink GR, Timmermann L. Impaired self-awareness of motor deficits in Parkinson's disease: association with motor asymmetry and motor phenotypes. Mov Disord. 2012 Sep 15;27(11):1443-7. doi: 10.1002/mds.25079. Epub 2012 Jun 18. PMID 22711290
- [Background] Clark JP, Adams SG, Dykstra AD, Moodie S, Jog M. Loudness perception and speech intensity control in Parkinson's disease. J Commun Disord. 2014 Sep-Oct;51:1-12. doi: 10.1016/j.jcomdis.2014.08.001. Epub 2014 Aug 23. PMID 25194745
- [Background] Carandini M, Churchland AK. Probing perceptual decisions in rodents. Nat Neurosci. 2013 Jul;16(7):824-31. doi: 10.1038/nn.3410. Epub 2013 Jun 25. PMID 23799475